CLINICAL TRIAL: NCT07063771
Title: The Safety and Efficacy of Irreversible Electroporation for the Treatment of Perivascular Liver Cancers
Brief Title: Safety and Clinical Efficacy of Histotripsy for Liver Cancers Adjacent to Major Intrahepatic Vessels
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202504040DIPB
Record Dates: First submitted 2025-06-12; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-06

CONDITIONS: Liver Tumors
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- treatment liver tumors (Experimental)
  Interventions: Device: Histotripsy

INTERVENTIONS:
Device: Histotripsy — Histotripsy is a tumor ablation technique developed in recent years that allows for non-invasive treatment of solid tumors using High-Intensity Focused Ultrasound (HIFU). This method works by physically focusing ultrasound energy at a single point within biological tissue, creating a focal zone of high-power, low-frequency ultrasound that induces mechanical fragmentation (histotripsy) and cavitation effects, dissolving the tissue into fragments and destroying tumor cells. Under real-time ultrasound imaging guidance, various scanning treatment protocols are used to move the focal point throughout the treatment zone, effectively ablating the tumor tissue. The destroyed tumor tissue is gradually absorbed by the body. Since this technique does not require needle puncture, electrode insertion, radiation, or thermal effects, it is minimally invasive and holds the potential to overcome the limitations of existing ablation technologies.

SUMMARY:
Malignant liver tumors are among the most common malignancies worldwide, with over 10,000 new cases diagnosed annually in Taiwan. Despite the variety of treatment options currently available for malignant liver tumors, the prognosis for patients with primary hepatocellular carcinoma or metastatic liver cancer remains disheartening. More than 8,000 people die from the disease each year. The majority of patients (approximately 70% to 85%) are diagnosed at an advanced stage or have tumors that are unresectable. In contrast, patients with smaller tumors have a much better chance of achieving a cure. Numerous studies have reported that patients who undergo hepatic lobectomy have a 5-year disease-free survival rate exceeding 50%. For tumors that are not surgically resectable, local ablation techniques such as Radiofrequency Ablation (RFA) have emerged as potentially curative alternatives. However, RFA has significant drawbacks: its percutaneous invasiveness can sometimes lead to bleeding or tumor seeding along the needle tract, and it may be less effective near blood vessels due to the heat-sink effect. Therefore, its application is currently limited to small liver tumors. Histotripsy is a tumor ablation technique developed in recent years that allows for non-invasive treatment of solid tumors using High-Intensity Focused Ultrasound (HIFU). This method works by physically focusing ultrasound energy at a single point within biological tissue, creating a focal zone of high-power, low-frequency ultrasound that induces mechanical fragmentation (histotripsy) and cavitation effects, dissolving the tissue into fragments and destroying tumor cells. Under real-time ultrasound imaging guidance, various scanning treatment protocols are used to move the focal point throughout the treatment zone, effectively ablating the tumor tissue. This clinical trial utilizes the Edison System, developed by HistoSonics Inc. (USA). The first multicenter Phase I human trial of this technology was conducted in 2018, lasting eight weeks and treating 11 patients with advanced, unresectable multifocal liver tumors. All targeted tumors were successfully ablated with no device-related adverse events. This research project aims to evaluate the clinical feasibility and advantages of this system in malignant liver tumor patients who are ineligible for surgical resection but are still candidates for local tumor ablation. To investigators plan to perform ablation under general anesthesia on 20 participants with liver tumors located within 1 cm of the inferior vena cava, hepatic veins, or bilateral portal vein trunks. Post-procedural complications will be monitored, and follow-up over 12 months will assess complete tumor ablation and intrahepatic recurrence to verify the system's clinical viability and potential benefits.

ELIGIBILITY:
Inclusion Criteria:

* Ages Eligible for Study: 18 Years and older
* Diagnosed with a malignant liver tumor at National Taiwan University Hospital. The diagnosis of liver cancer was based on the international diagnostic criteria of the AASLD, while the diagnosis of other primary malignant liver tumors and metastatic liver tumor was based on pathological diagnostic standards
* Unsuitable for surgical resection. the tumor is located less than 1 cm from critical vascular structures, including the inferior vena cava, hepatic veins, and both main branches of the portal vein.
* Have at least one, but less than or equal to 3 tumors, At least one of them met the third criterion
* Each tumor must be ≤ 5 cm in diameter,
* Child-Pugh class A-B,
* Eastern Cooperative Oncology Group (ECOG) score of 0-1,
* American Society of Anesthesiologists (ASA) score ≤ 3,
* Adequate bone marrow and liver function (1). Platelet count ≥ 100 K/Μl(2). Total bilirubin ≦ 2.5 mg/dL(3). ALT and AST < 5 x upper limit of normal (4). PT-INR ≦ 2.0.
* Prior Informed Consent Form
* Life expectancy of at least 3 months.
* Maximum tumor depth ≤14 cm from the skin surface
* Patients who are in good physical condition and able to tolerate endotracheal intubation and general anesthesia

Exclusion Criteria:

* Women who are pregnant or women of child-bearing potential who are not using an acceptable method of contraception,
* Received treatment with an investigational agent/ procedure within 30 days prior to Histotripsy treatment
* Acute infection or inflammation, acute and severe dysfunction of heart, liver and kidney.
* Known history of HIV infection
* Tumor not clearly visualized on ultrasound
* No safe ultrasound pathway due to scarring, bowel gas, calcified tumor, or bone interference
* Prior radiotherapy within 30 days before or after treatment
* Arterial calcification in the treatment area
* Investigator-assessed contraindications
* Inability to undergo CT/MRI imaging
* Severe anesthesia intolerance
* Tumor invasion of major vessels, gastrointestinal tract, or respiratory tract

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of SF-36 and VAS with preoperative baseline within six months | six months
  The main goals are to confirm if the quality of life of subjects improves after treatment with a focused ultrasound system and to assess the safety of the treatment. The acceptable safety range, according to CTCAE Version 5.0 criteria, should be Grade 3 or below.

SECONDARY OUTCOMES:
Comparison of Tumor Volume Before and After Treatment | 12 months
  Using CT/MRI images to assess changes in tumor volume before and after focused ultrasound treatment, and the RECIST (Response Evaluation Criteria in Solid Tumors) criteria are commonly applied.